CLINICAL TRIAL: NCT04949438
Title: A Single Dose, Non-Randomised, Open-Label, Parallel Group Study to Assess the Pharmacokinetics, Safety and Tolerability of AZD4831 in Participants With Severe Renal Impairment and Healthy Volunteers
Brief Title: A Study to Assess the Pharmacokinetics (Uptake of Drugs by the Body), Safety and Tolerability of AZD4831 in Participants With Severe Renal Impairment and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6580C00009
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Renal Impairment
Keywords: AZD4831; Pharmacokinetics; Estimated glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency | interventions — AZD4831

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Participants with severe renal impairment (Experimental): Participants with severe renal impairment will receive a single oral dose of AZD4831 on Day 1.
  Interventions: Drug: AZD4831
- Cohort 2 :Healthy participants (Experimental): Healthy participants will receive a single oral dose of AZD4831 on Day 1.
  Interventions: Drug: AZD4831

INTERVENTIONS:
Drug: AZD4831 — Participants will receive a single dose of AZD4831 administered with 240 mL of water after an overnight fast of at least 10 hours.

SUMMARY:
This is a study to compare AZD4831 pharmacokinetic (PK) parameters between participants with severe renal impairment and matched healthy volunteers following a single dose administration.

DETAILED DESCRIPTION:
All participants will receive a single oral dose of AZD4831 under fasted conditions and will be involved in the study approximately 2 weeks after dosing and up to approximately 38 days from screening.

Approximately 10 participants will be enrolled into each of the 2 cohorts parallelly and receive the study intervention to achieve 8 evaluable participants in each cohort.

* Cohort 1: 10 participants with severe renal impairment (Estimated glomerular filtration rate [eGFR] of ≥15 to <30 mL/min/1.73m^2)
* Cohort 2: 10 matched healthy volunteers with normal renal function (eGFR of ≥90 mL/min/1.73m^2).

The study will comprise of the following study periods:

* Screening period (21 days): participants will be screened for eligibility.
* Treatment period (3 days): participants will be admitted to the study centre in the evening of (Day -1) the day before administration of a single oral dose of AZD4831 (Day 1), and will be discharged after at least 24 h post-dose (Day 2).
* Follow-up period (13±2 days): participants will attend 5 visits at the study centre for PK sampling and safety assessments on Days 3, 5, 8, 11 and 15.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be 18 to 80 (inclusive) years of age, at the time of signing the informed consent.
* The age of participants in Cohort 2 (matched healthy volunteers) must not be lesser than 10 years below the lowest age in Cohort 1 (participants with severe renal impairment) or greater than 10 years above the highest age in Cohort 1.

Healthy volunteers only (Cohort 2):

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* An eGFR of ≥90 mL/min/1.73m^2 as determined at screening using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.

Participants with severe renal impairment only (Cohort 1):

* An eGFR of ≥15 to <30 mL/min/1.73m^2 as determined at screening using the CKD-EPI formula.
* Stable renal function.
* If participants are on statin, ACEi/ARB, beta-blocker, diuretic or on any other cardiorenal relevant treatment, the dose should be stable at least 2 weeks prior to screening (Visit 1).
* Body weight of at least 50 kg and body mass index (BMI) within the range ≥18 to ≤35 kg/m^2.
* BMI of participants in Cohort 2 (healthy volunteers) must not be more than 20% below the lowest BMI in Cohort 1 (participants with severe renal impairment) or more than 20% above the highest BMI in Cohort 1.
* Male or female of non-childbearing potential.
* There should be an equal number of male and female participants in Cohort 2 (healthy volunteers) as in Cohort 1 (participants with severe renal impairment).

  1. Male participants: All male participants should use methods of contraception consistent with local regulations for those participating in clinical studies.
  2. Highly effective birth control methods are defined as those that can achieve a failure rate of less than 1% per year when used consistently and correctly
  3. Female participants: Must have a negative serum pregnancy test at screening and admission to the study centre (Day -1), must not be lactating and must be of non-childbearing potential confirmed at screening.
* Male participants should not donate sperm for the duration of the study and for at least 90 days after the last study follow-up visit.
* Provision of signed and dated written Optional Genetic Research Information informed consent prior to collection of samples for optional genetic research.

Exclusion Criteria:

* Any evidence of a clinically significant disease or disorder.
* Positive hepatitis C antibody, hepatitis B virus surface antigen, hepatitis B virus core antibody, or human immunodeficiency virus I or II at screening (Visit 1).
* History of drug or alcohol abuse within 1 year of screening or positive test for drugs of abuse and alcohol at screening and admission to the study centre.
* History of allergy/hypersensitivity to drugs with a similar chemical structure or class to AZD4831or any of the excipients of the product.
* Any of the following signs or confirmation of Corona Virus 2019 (COVID-19) infection

  a. Participant has a positive severe acute respiratory syndrome coronavirus 2 reverse transcription-polymerase chain reaction test result within 2 weeks before screening (Visit 1) or between screening and admission to study centre (Visit 2).

  (i) Clinical signs and symptoms consistent with COVID-19 (eg, fever, dry cough, dyspnoea, sore throat, fatigue) 2 weeks before screening (Visit 1) or between screening and admission to study centre (Visit 2).

(ii) Participant has been previously hospitalised with COVID-19 infection within the last 3 months.

Healthy volunteers only (Cohort 2):

- History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.

Participants with severe renal impairment only (Cohort 1):

* Renal transplant participants or participants on dialysis.
* Use of concurrent medication, which affect creatinine clearance such as cephalosporin antibiotics, ascorbic acid, trimethoprim, cimetidine, or quinine within days of admission to the study centre (Day -1).
* Use of drugs with enzyme-inducing properties such as St John's Wort within 7 days or 5 half-lives (whichever is longer) prior to screening (Visit 1).
* Any concomitant medications known to be associated with Torsades de Pointes or strong cytochrome P450 3A4 (CYP3A4) inducers or inhibitors.

Healthy volunteers only (Cohort 2):

- Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol), herbal remedies, megadose vitamins and minerals within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the study intervention and until completion of the follow-up visits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | From Day 1 to Day 15
  Assessment of Cmax of a single oral dose of AZD4831 in participants with severe renal impairment compared with that in matched healthy volunteers.
Time to reach maximum observed plasma concentration (tmax) | From Day 1 to Day 15
  Assessment of tmax of a single oral dose of AZD4831 in participants with severe renal impairment compared with that in matched healthy volunteers.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½λz) | From Day 1 to Day 15
  Assessment of t½λz of a single oral dose of AZD4831 in participants with severe renal impairment compared with that in matched healthy volunteers.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | From Day 1 to Day 15
  Assessment of CL/F of a single oral dose of AZD4831 in participants with severe renal impairment compared with that in matched healthy volunteers.
Apparent total non-renal body clearance of drug from plasma after extravascular administration (CLNR/F) | From Day 1 to Day 15
  Assessment of CLNR/F of a single oral dose of AZD4831 in participants with severe renal impairment compared with that in matched healthy volunteers.
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | From Day 1 to Day 15
  Assessment of Vz/F of a single oral dose of AZD4831 in participants with severe renal impairment compared with that in matched healthy volunteers.
Area under the plasma concentration-curve from time zero to time of last quantifiable concentration (AUClast) | From Day 1 to Day 15
  Assessment of AUClast of a single oral dose of AZD4831 in participants with severe renal impairment compared with that in matched healthy volunteers.
Area under plasma concentration-time curve from time zero to infinity (AUCinf) | From Day 1 to Day 15
  Assessment of AUCinf of a single oral dose of AZD4831 in participants with severe renal impairment compared with that in matched healthy volunteers.
Renal clearance of drug from plasma (CLR) | Days 1 and 2
  Assessment of CLR of a single oral dose of AZD4831 in participants with severe renal impairment compared with that in matched healthy volunteers.

SECONDARY OUTCOMES:
Number of participants with adverse events | From Screening (Day -21 to Day -1) until Day 15 or Early Termination Visit
  Assessment of the safety and tolerability of a single oral dose administration of AZD4831 in participants with severe renal impairment and their matched healthy volunteers.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home